CLINICAL TRIAL: NCT00824590
Title: A Phase 1, Non-Randomized, Open-Label, Single-Dose Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Dimebon [PF 01913539] In Subjects With Severely-Impaired And Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1451019
Record Dates: First submitted 2009-01-12; First posted 2009-01-19 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: Dimebon; renal impairment; pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease; Renal Insufficiency | interventions — latrepirdine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe renal impairment group (Experimental): Subjects with severe renal impairment defined by creatinine clearance of less than 30 mL/min but not yet on dialysis
  Interventions: Drug: Dimebon
- normal renal function (Experimental): Subjects with normal renal function defined by creatinine clearance of greater than 80 mL/min and demographically comparable to subjects with impaired renal function
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — a single oral dose of 20 mg Dimebon
  Arms: Severe renal impairment group
Drug: Dimebon — a single oral dose of 20 mg Dimebon
  Arms: normal renal function

SUMMARY:
This study is to compare the pharmacokinetics of Dimebon in subjects with severe renal impairment to subjects with normal renal function after oral administration of a single oral 20-mg dose of Dimebon. This study is also to assess the safety and tolerability of a single oral 20-mg dose of Dimebon in subjects with severe renal impairment and subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 18 and 75 years, inclusive
* For severe renal impairment group, subjects with creatinine clearance of less than 30 mL/min, but not yet on dialysis and in good general health commensurate with the population with chronic renal disease; however, subjects with type 1 and 2 diabetes that are reasonably controlled and who do not have a predisposition to severe hypoglycemia can both be included.
* For normal renal function group, healthy subjects with creatinine clearance of greater than 80mL/min and demographically comparable to subjects with impaired renal function

Exclusion Criteria:

* Pregnant or nursing women; women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to the first dose of study medication.
* For normal renal function group, use of prescription or non-prescription drugs, vitamins, or dietary supplements within 7 days of 5 half-lives (whichever is longer) prior to the first dose of study medication.

Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. Acetaminophen at doses of ≤ 2 grams/day is permitted.

* For renal impairment group, a known history of clinically significant coronary heart disease, cerebrovascular disease or peripheral vascular disease and/or an event/intervention during the past 6 months. Systemic therapy with CYP3A or CYP2D6 inhibitors within 7 days or 5 halflives (whichever is longer) prior to the first dose of trial medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentrations | 96

SECONDARY OUTCOMES:
Safety assessment including physical/neurological examination findings, clinical safety laboratory assessments, 12-lead ECGs, vital sign measurements, and adverse event monitoring. | 96

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Saint Paul, Minnesota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451019&StudyName=A%20Phase%201%2C%20Non-Randomized%2C%20Open-Label%2C%20Single-Dose%20Study%20To%20Evaluate%20The%20Pharmacokinetics%2C%20Safety%2C%20And%20Tolerability%20Of%20Dimebon%20%5BPF